CLINICAL TRIAL: NCT03309488
Title: Basophil Activation Test to Diagnose Food Allergy
Acronym: BAT2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 197886
Record Dates: First submitted 2017-07-07; First posted 2017-10-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Food Allergy; Food Allergy in Infants; Food Allergy in Children; Food Allergen Sensitisation; Milk Allergy; Egg Allergy; Nut Allergy
Keywords: Food allergy; Milk allergy; Egg allergy; Nut allergy; Basophil activation test; Diagnosis; Specific IgE; Skin prick test
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Nut Hypersensitivity; Disease | interventions — Basophil Degranulation Test; Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Food allergic: Patients with a positive oral challenge to the food being studied.
  Interventions: Diagnostic Test: Oral food challenge
- Non food allergic: Patients with a negative oral challenge to the food being studied.
  Interventions: Diagnostic Test: Oral food challenge

INTERVENTIONS:
Diagnostic Test: Oral food challenge — Patients with suspected food allergy will undergo clinical and dietary assessments and oral food challenge. Different allergy tests will be performed, including skin prick test, specific IgE test and basophil activation test, and its diagnostic utility will be determined against the clinical gold-standard.
  Other Names: Basophil activation test; Skin prick test; Specific IgE test

SUMMARY:
The BAT II Study is a cross-sectional diagnostic study in which children with suspected IgE-mediated allergy to foods (namely cow's milk, egg, sesame and cashew), as defined by a history of an immediate-type allergic reaction to a food or no history of food consumption or the presence of food-specific IgE as documented by skin prick test or serum specific IgE, will undergo a diagnostic work-up to confirm or refute the diagnosis of IgE-mediated food allergy. Participants will be prospectively recruited from specialised Paediatric Allergy clinics in London and will undergo skin prick testing (SPT), specific IgE testing to allergen extracts and allergen components, basophil activation test (BAT) and oral food challenge. The diagnostic accuracy of the BAT and of other allergy tests will be assessed against the clinical gold-standard.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥6 months and <16 years old;
2. Suspected IgE-mediated food allergy defined by:

   * History of an immediate-type allergic reaction to a specific food or
   * No history of consumption of the specific food or
   * IgE sensitisation documented by skin prick test (≥1 mm) or serum specific IgE (≥0.10 KU/L);
3. Avoidance of the specific food for at least 2 days prior to blood collection for BAT and specific IgE and prior to the challenge;
4. Informed consent obtained from parent or guardian and assent obtained from the child.

Exclusion Criteria:

1. Clinically significant chronic illness other than atopic diseases;
2. Previous history of severe life-threatening reaction to the suspected food with documented decrease in oxygen saturation (<90%), hypotension (≥20% reduction in systolic blood pressure) and/or admission to intensive care;
3. Unwillingness to comply with study procedures, namely to undergo a diagnostic food challenge;
4. Contra-indication for diagnostic food challenge, namely:

   * Uncontrolled atopic diseases (e.g. eczema, asthma, rhinitis);
   * Chronic medical conditions that pose significant risk in the event of anaphylaxis or treatment of anaphylaxis (e.g. cardiac disease, severe lung disease, pregnancy, mastocytosis);
   * Inability to discontinue medications that might interfere with assessment or safety (e.g. antihistamines, β-agonists, β-blockers, NSAIDs, ACE inhibitor, antacids);
   * Recent (within 7-14 days) treatment with systemic steroids or prolonged high-dose systemic steroids or immunosuppressants;
5. Undergoing treatment with omalizumab, food allergen immunotherapy or other systemic immunomodulatory treatment;
6. Inability to stop anti-histamines prior to SPT.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children seen in specialized Pediatric Allergy clinics with suspected allergy to one of the foods studied, namely milk, egg, sesame and nuts.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the basophil activation test (for each individual food allergy) | 3 years
  Accuracy of %CD63+ basophils

SECONDARY OUTCOMES:
Diagnostic accuracy of SPT, specific IgE to extracts and to single allergens | 3 years
  Accuracy of weal diameter or level of IgE
Association between BAT and severity of symptoms during challenges | 3 years
  Correlation between %CD63+ basophils and severity grade
Association between BAT and threshold of reactivity during challenges | 3 years
  Correlation between CD-sens and cumulative threshold dose

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Santos, MD PhD, Principal Investigator — King's College London
Locations (1):
- Pediatric Allergy Clinical Research Facility, Evelina Children's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bartha I, Boyd H, Foong RX, Krawiec M, Marques-Mejias A, Marshall HF, Radulovic S, Harrison F, Antoneria G, Jama Z, Kwok M, Pietraszewicz E, Eghleilib M, Ricci C, Marrs T, Lack G, Du Toit G, Santos AF. The Basophil Activation Test Is the Most Accurate Test in Predicting Allergic Reactions to Baked and Fresh Cow's Milk During Oral Food Challenges. Allergy. 2025 Oct;80(10):2861-2873. doi: 10.1111/all.16675. Epub 2025 Aug 13. PMID 40808324
- [Derived] Marques-Mejias A, Radulovic S, Foong RX, Bartha I, Krawiec M, Kwok M, Jama Z, Harrison F, Ricci C, Lack G, Du Toit G, Santos AF. Partial Egg Consumption Modifies the Diagnostic Performance of Allergy Tests to Predict Outcome of Double-Blind Placebo-Controlled Food Challenges to Egg. J Allergy Clin Immunol Pract. 2024 Mar;12(3):660-669.e5. doi: 10.1016/j.jaip.2023.12.036. Epub 2023 Dec 27. PMID 38157981